CLINICAL TRIAL: NCT00718081
Title: A Multicenter, Randomized, Placebo-Controlled Phase 2 Study to Evaluate the Clinical Efficacy, Safety, and Tolerability of ARX-F01 Sublingual Sufentanil in Patients Undergoing Major Abdominal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARX-C-005
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-12

CONDITIONS: Major Upper or Lower Abdominal Surgery
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Oral Sufentanil
  Interventions: Drug: Oral sufentanil
- 2 (Experimental): Oral sufentanil
  Interventions: Drug: Oral sufentanil
- 3 (Placebo Comparator): Oral dosage of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral sufentanil — Oral dosage of sufentanil
  Arms: 1; 2
Drug: Placebo — Oral dosage of placebo
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate dosages of ARX-F01 (opioid pain medication) versus a placebo (or sugar pill) for the treatment of post-operative pain in subjects following abdominal surgery. We hypothesize that subjects receiving placebo will have poor pain relief and will drop out of the study sooner and more often than the ARX-F01 treated subjects.

ELIGIBILITY:
Inclusion Criteria at Screening:

1. Male or female patients between 18 to 80 years of age.
2. Patient is scheduled to undergo an upper or lower abdominal surgery under general anesthesia.
3. Patient must be classified as American Society of Anesthesiologists (ASA) class I - III.
4. Patient must have Body Mass Index [BMI = weight (kg)/height (m2)] between 18 and 39, inclusively.
5. Female patients of childbearing potential must be using an effective method of birth control from the screening visit through the end of study. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or postmenopausal for ≥1 year, must be specified in the patient's case report form (CRF).
6. The patient must be willing and able to understand the study procedures and the use of pain scales, and to communicate meaningfully with the study personnel.
7. The patient must provide written informed consent and sign the Informed Consent

Exclusion Criteria at Screening:

1. Patient is scheduled to undergo a laparoscopically-assisted abdominal surgery.
2. Patient has previously not responded to opioid analgesics for treatment of pain.
3. Patient is currently taking or has taken an opioid for more than 30 consecutive days of daily use at a daily dose equivalent to greater than 15 mg morphine within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
4. Patient has an allergy or hypersensitivity to opioids.
5. Patient currently has sleep apnea that has been documented by a sleep laboratory study.
6. Patient has any screening laboratory test value outside the laboratory normal range which is considered clinically significant by the Investigator.
7. Patient is a woman who is pregnant or lactating.
8. Patient has psychiatric disease or encephalopathy severe enough to prevent patient from providing reliable study documentation.
9. Patient, in the Investigator's judgment, does not have adequate ability to read and understand English.
10. Patient has a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including chronic abdominal pain or active infection.
11. Patient has clinically significant renal or liver impairment which could affect metabolism or clearance of sufentanil.
12. Patient has a painful physical condition other than acute abdominal pain that, in the opinion of the Investigator, may confound post-operative pain assessments.
13. Patient has a history of drug, prescription medicine, or alcohol abuse within the past 2 years or a positive drug screen test for cocaine, amphetamines, barbiturates, phencyclidine, or methadone at screening.
14. Patient is receiving oxygen therapy at the time of screening.
15. Patient has participated in a clinical trial of an investigational drug or device within 30 days of screening visit or is scheduled to receive an investigational product other than ARX-F01 while participating in this study.

Exclusion Criteria at Randomization (during early PACU time period):

1. Patient has a respiratory rate that is less than 8 breaths per minute or greater than 24 breaths per minute.
2. Patient has arterial oxygen saturation by pulse oximetry (SpO2) of less than 90% with supplemental oxygen.
3. Patient is not able to answer questions and follow commands.
4. Patient has vomiting that is not responsive to standard treatment.
5. The surgical procedure from incision to closure was longer than 4 hours.
6. There have been any deviations from the surgical or anesthetic protocols as specified in Section 6.1.2.1.

approved by the Institutional Review Board (IRB).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Trio Clinical Research, Durham, North Carolina, United States

REFERENCES:
- [Result] Minkowitz HS, Singla NK, Evashenk MA, Hwang SS, Chiang YK, Hamel LG, Palmer PP. Pharmacokinetics of sublingual sufentanil tablets and efficacy and safety in the management of postoperative pain. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):131-9. doi: 10.1097/AAP.0b013e3182791157. PMID 23271030

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil NanoTab 10 mcg | Sufentanil NanoTab 15 mcg | Placebo NanoTab
Started | 29 | 29 | 30
Completed | 22 | 25 | 9
Not Completed | 7 | 4 | 21
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lack of Efficacy | 7 | 3 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil NanoTab 10 mcg | Sufentanil NanoTab 15 mcg | Placebo NanoTab | Total
Number analyzed (Participants) | 29 | 29 | 30 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 28 | 80
  >=65 years | 3 | 3 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.7) | 45.3 (11.3) | 46.8 (10.1) | 46.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 28 | 84
  Male | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 30 | 88

OUTCOME MEASURES:

1. Primary Outcome: SPID-12
Description: The primary outcome measure is the summed pain intensity difference over the 12-hour study period (SPID-12). A pain intensity score ranging from 0 (no pain) to 10 (worst possible pain) is obtained at baseline and throughout the 12 hour study period. The SPID-12 is calculated by summing the difference between baseline pain score and pain score at each assessment time point. The scores after summing could range from -122 to +122. A higher SPID-12 score is better.
Time Frame: 12 hours after surgery
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil NanoTab 10 mcg | Sufentanil NanoTab 15 mcg | Placebo NanoTab
Number analyzed (Participants) | 29 | 29 | 30
units on a scale | 22.41 (3.61) | 27.56 (3.50) | 2.93 (3.46)
Statistical Analysis 1: Comparison: Sufentanil NanoTab 10 mcg vs Placebo NanoTab; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 19.48, Standard Error of Mean 4.92
Statistical Analysis 2: Comparison: Sufentanil NanoTab 15 mcg vs Placebo NanoTab; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 24.62, Standard Error of Mean 4.86

2. Secondary Outcome: Proportion of Patients Who Responded Very Good or Excellent in Patient Global Evaluation of Pain Relief
Description: At the end of the 12-hour study period each patient rated their overall pain relief since starting study drug on a 5-point scale: poor, fair, good, very good or excellent.
Time Frame: Up to 12 hours after surgery
Measure: Number; unit: percentage of patients
Arm/Group | Sufentanil NanoTab 10 mcg | Sufentanil NanoTab 15 mcg | Placebo NanoTab
Number analyzed (Participants) | 29 | 29 | 30
percentage of patients | 38 | 55 | 10

ADVERSE EVENTS:
Arm/Group | Sufentanil NanoTab 10 mcg | Sufentanil NanoTab 15 mcg | Placebo NanoTab
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 15/29 | 17/29 | 15/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab 10 mcg (N=29) | Sufentanil NanoTab 15 mcg (N=29) | Placebo NanoTab (N=30)
dizziness (Nervous system disorders) | 1 | 0 | 1
headache (Nervous system disorders) | 2 | 1 | 2
insomnia (Psychiatric disorders) | 1 | 1 | 0
nausea (Gastrointestinal disorders) | 13 | 14 | 12
pruritus (Skin and subcutaneous tissue disorders) | 2 | 5 | 1
pyrexia (General disorders) | 0 | 0 | 1
vomiting (Gastrointestinal disorders) | 2 | 0 | 2
abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 — All adverse events in this table were assessed by the PI as possibly or probably related to study drug
hypothermia (General disorders) | 0 | 0 | 1
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
requires prior consent